CLINICAL TRIAL: NCT05740852
Title: Analysis of Risk Factors of Postoperative Pulmonary Infection in Patients With Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XijingHCJF
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-01

CONDITIONS: Esophageal Neoplasms; Pneumonia
MeSH Terms: conditions — Esophageal Neoplasms; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infection: Patients who developed pulmonary infection after radical resection of tumor
- Without infection: Patients without pulmonary infection after radical resection of tumor

SUMMARY:
The goal of this observational study is to learn about in describe participant population. The main questions it aims to answer are:

* What are the risk factors of postoperative pulmonary infection in patients with esophageal cancer？
* Whether we could establish a clinical prediction model to provide basis for early clinical intervention or not? Participants will describe the main tasks participants will be asked to do, treatments they'll be given and use bullets if it is more than 2 items. If there is a comparison group: Researchers will compare insert groups to see if insert effects.

DETAILED DESCRIPTION:
Data were collected from the electronic medical records of Xijing Hospital. Each record is entered by two team members working simultaneously to ensure data accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of esophageal cancer;
* Radical resection of tumor for the first time;
* No distant metastasis was observed in preoperative examination

Exclusion Criteria:

* Patients with preoperative pulmonary infection or symptoms of pulmonary infection;
* Patients with tracheal intubation assisted ventilation before surgery;
* Patients with preoperative lung imaging changes or abnormal white blood cells in blood routine;
* Patients undergoing emergency surgery;
* Patients with other cancers;
* Patients with incomplete clinical data.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2016 to December 2021, patients with esophageal cancer were hospitalized for surgery in the Department of Gastroenterology, Xijing Hospital.
Sampling Method: Probability Sample
Enrollment: 1688 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Pneumonia | A week after radical resection of tumor
  Pulmonary infection in patients with esophageal cancer after radical resection of tumor